CLINICAL TRIAL: NCT06728085
Title: A Pragmatic Trial on Actions For Collaborative Community Engaged Strategies for HPV
Acronym: ACCESS-HPV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Nigerian Institute of Medical Research (Other Government); University of North Carolina, Chapel Hill (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 20240291; R01CA271033 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-12-11 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: HPV
Keywords: HPV Vaccination; HPV Screening

STUDY DESIGN:
Intervention Model Description: Hybrid Type II, stepped-wedge cluster randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mother-Daughter Day HPV Campaign (Experimental): Each of the 18 local government areas begin as part of the control condition and are block-randomized into four waves in the pre-implementation phase, with each wave beginning 2 months after the start of the prior wave and lasting for 6 months. The local government areas will implement the intervention for 6 months, followed by a post implementation phase.
  Interventions: Behavioral: Baseline Assessment For Mother-Daughter Day HPV Campaign; Behavioral: Implement Mother-Daugther Day HPV Campaign; Behavioral: Post-Implementation Follow-Up

INTERVENTIONS:
Behavioral: Baseline Assessment For Mother-Daughter Day HPV Campaign — Pre-Implementation:
  Identify, screen, and enroll mother-daughter dyads in the study to participate in the upcoming Mother-Daughter Day event on HPV vaccination and screening.
  Complete baseline surveys with enrolled participants. Distribute reminder cards and send text messages to mother-daughter dyads who agree to participate in the mother-daughter day campaign.
  Other Names: Pre-Implementation Phase
Behavioral: Implement Mother-Daugther Day HPV Campaign — Tailor and adapt to context: Mother-Daughter Day campaigns will be tailored and adapted to the local contexts within the 18 LGA.
  Trained community health workers will implement the tailored Mother-Daughter Campaign by providing education on cervical cancer control and educational materials on HPV vaccination and HPV screening.
  Engage mothers and daughters with on-site access to services: This includes offer of onsite vaccinations to girls by study nurse as well as offer of onsite self-collection screening kits to mothers and caregivers in a private area, along with instructions on how to use and return the sample.
  Distribute gift bags with HPV vaccination cards, follow-up reminders, and linkage cards for participants with positive test results, as community health workers continue to provide onsite support and assistance.
  Other Names: Implementation Phase
Behavioral: Post-Implementation Follow-Up — A follow-up invitation will be sent to participate in a consultative phone call with study health workers to review self-collection results.
  Participants with positive HPV test results will be linked to follow-up care and treatment.
  Other Names: Post-Implementation Phase

SUMMARY:
The present study expands on the investigators' earlier pilot study, outlined in ClinicalTrial ID#: NCT06010108. The Actions for Collaborative Community-Engaged Strategies for HPV (ACCESS-HPV), locally referred to as 4 Girls and Women (4GW) in Nigeria, seek to utilize a participatory crowdsourcing approach to enhance HPV prevention efforts among mother-daughter dyads. Specifically, the investigators aim to 1) develop a new combined HPV vaccination and HPV self-collection campaign for mothers/daughters using crowdsourcing open calls and learning community groups, 2) determine whether the co-developed final combined crowdsourced campaign will increase HPV vaccination rates among girls and promote HPV self-collection among mothers, and 3) estimate the impact and cost-effectiveness of the combined crowdsourced campaign in Nigeria.

DETAILED DESCRIPTION:
Following the completion of the open contests, designathons and boot-camp training, seven trained teams (with seven distinct interventions) were selected to undergo a 6-month pilot assessment in the community. Preliminary findings from the feasibility study suggest that crowdsourced interventions have the potential to impact uptake of HPV vaccinations among girls and HPV screening among mothers in Nigeria. As a result, the investigators identified key components from the top 2 interventions to form a single intervention that will be evaluated in the next phase of the research. Thus, the current protocol is focused on evaluating the effectiveness of a combined, crowdsourced intervention on HPV vaccination among girls and HPV screening among mothers in Nigeria.

Using a hybrid effectiveness-implementation type II pragmatic stepped-wedge cluster randomized control trial, this study will test the effectiveness of an implementation strategy bundle; a crowdsourced, tailored, community-engaged, mother-daughter HPV campaign on increasing uptake of HPV vaccination among girls aged 9-14 and HPV screening uptake among women aged 30-65 in Nigeria. The mother-daughter campaign will be tailored to local sites and conducted among 612 mother-daughter dyads (1,224 participants) recruited from 18 LGAs in six geopolitical zones of Nigeria. Upon enrollment, trained community health workers (two per LGA) will collect baseline data, and implement a mother-daughter day campaign that will provide education on cervical cancer control and access to onsite services for HPV vaccination and screening in a private area and engage mothers and daughters simultaneously to increase uptake of the services. A mixed-methods evaluative and iterative assessment will be conducted using Proctor's Implementation Outcomes Framework and the PEN-3 cultural model. The primary outcomes are the uptake of HPV preventive measures -HPV vaccination (one dose) among girls (ascertained by on-site records of vaccine uptake) and HPV self-collection completion among mothers (ascertained by laboratory receipt of self-collected specimens) within 6-months of trial enrollment. Pre-post effectiveness and cost of study components are embedded in the implementation and sustainment phases, with comparison to pre-implementation data assessed for each LGA.

ELIGIBILITY:
Inclusion Criteria:

* Female participants
* Aged between 9 and 14 years old for girls/daughters
* Aged between 30 and 65 years old for mothers (mothers defined as any female caregiver, including biological and surrogate mothers or close relatives who meet the eligibility criteria)
* Residing and planning to reside in any of the 18 local government areas for the next 12 months and willing to participate
* Girls must be unvaccinated for HPV.
* Mother must have no recent (at least within 5 years cervical cancer screening)
* Mothers or caregivers must own a mobile phone to follow up with both daughters and mothers.
* Participants must agree to the informed consent in English before enrolling in the study.

Exclusion Criteria:

* Inability to comply with the study protocol
* Recently vaccinated girls for HPV
* Recently screened mothers for HPV within the last 5 years
* Illness, cognitive impairment, or threatening behavior with acute risk to self or others
* No informed consent or cell phone

Ages: 9 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female participants
Enrollment: 1838 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Uptake of HPV Vaccination among girls/daughters | Up to 6 months of enrollment
  The proportion of eligible girls who receive at least one dose of HPV vaccine. This will be ascertained by documentation on HPV vaccination cards
Uptake of HPV Self-collection among mothers/caregivers | Up to 6 months of enrollment
  The proportion of eligible women who complete an HPV self-collection. This will be ascertained by laboratory receipt of self-collected specimens.

SECONDARY OUTCOMES:
Intervention Acceptability | Measured at baseline, 3 months, and 6 months.
  This will be measured using the Acceptability of Intervention Measure (AIM). The subscale is evaluated using a 5-point Likert scale, ranging from 1 to 5, with higher scores reflecting higher levels of acceptability. Cronbach alpha=0.85
Intervention Appropriateness | Measured at baseline, 3 months, and 6 months.
  This will be assessed using the Intervention Appropriateness Measure (IAM). The subscale is evaluated using a 5-point Likert scale, ranging from 1 to 5, with higher scores indicating higher levels of appropriateness. Cronbach alpha=0.91
Intervention Feasibility | Measured at baseline, 3 months, and 6 months.
  This will be assessed using the Feasibility of Intervention Measure (FIM). The subscale is rated on a 5-point Likert scale, 1 to 5, with higher scores indicating higher levels of feasibility.
Penetration (i.e., population dose) | Measured at baseline, 3 months, and 6 months.
  The extent to which components of the mother-daughter HPV campaigns are institutionalized within participating local government area.
Implementation Fidelity | Measured at baseline, 3 months, and 6 months.
  This will be assessed both quantitatively and qualitatively using the following four dimensions: (1) Frequency: number of intervention-related interactions; (2) Duration: length of each component of the intervention; (3) Content: the knowledge or behavioural change the combined intervention seeks to deliver to the mother/daughter dyads; and (4) Coverage: the number of mother/daughter dyads who receive the intervention as intended over the number of participants who are enrolled.
Sustainment | Measured at baseline, 3 months, 6 months, and 12 months
  Measured using the Sustainment Measurement System Scale. Items will be rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (all the time), with lower scores indicating lower levels of agreement while higher scores indicating higher levels of agreement.

OTHER OUTCOMES:
Key Implementation Factors | Up to 12 months of follow-up
  Guided by the RE-AIM framework for implementation science, semi-structured, in-depth interviews will be conducted at the individual and setting levels to explore the factors associated with the implementation of the intervention (e.g., reach, adoption, implementation, and maintenance).

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Iwelunmor, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Nigerian Institute of Medical Research, Yaba, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kpokiri EE, Wapmuk A, Obiezu-Umeh C, Nwaozuru U, Gbaja-Biamila T, Obionu I, Kokelu E, Smith J, Benedict AN, Ajenifuja K, Babatunde AO, Ezechi O, Tucker JD, Iwelunmor J. A designathon to co-create HPV screening and vaccination approaches for mothers and daughters in Nigeria: findings from a community-led participatory event. Res Sq [Preprint]. 2024 Jan 29:rs.3.rs-3829727. doi: 10.21203/rs.3.rs-3829727/v1. PMID 38352305
- [Background] Cates JR, Shafer A, Diehl SJ, Deal AM. Evaluating a County-Sponsored Social Marketing Campaign to Increase Mothers' Initiation of HPV Vaccine for their Pre-teen Daughters in a Primarily Rural Area. Soc Mar Q. 2011 Spring;17(1):4-26. doi: 10.1080/15245004.2010.546943. PMID 21804767
- [Background] Lee H, Kim M, Cooley ME, Kiang PN, Kim D, Tang S, Shi L, Thiem L, Kan P, Peou S, Touch C, Chea P, Allison J. Using narrative intervention for HPV vaccine behavior change among Khmer mothers and daughters: A pilot RCT to examine feasibility, acceptability, and preliminary effectiveness. Appl Nurs Res. 2018 Apr;40:51-60. doi: 10.1016/j.apnr.2017.12.008. Epub 2017 Dec 18. PMID 29579499
- [Background] Scarinci IC, Hansen B, Kim YI. HPV vaccine uptake among daughters of Latinx immigrant mothers: Findings from a cluster randomized controlled trial of a community-based, culturally relevant intervention. Vaccine. 2020 May 22;38(25):4125-4134. doi: 10.1016/j.vaccine.2020.03.052. Epub 2020 Apr 27. PMID 32354671
- [Background] Winer RL, Gonzales AA, Noonan CJ, Buchwald DS. A Cluster-Randomized Trial to Evaluate a Mother-Daughter Dyadic Educational Intervention for Increasing HPV Vaccination Coverage in American Indian Girls. J Community Health. 2016 Apr;41(2):274-81. doi: 10.1007/s10900-015-0093-2. PMID 26399648
- [Background] Abuelo CE, Levinson KL, Salmeron J, Sologuren CV, Fernandez MJ, Belinson JL. The Peru Cervical Cancer Screening Study (PERCAPS): the design and implementation of a mother/daughter screen, treat, and vaccinate program in the Peruvian jungle. J Community Health. 2014 Jun;39(3):409-15. doi: 10.1007/s10900-013-9786-6. PMID 24276617
- [Background] Amponsah-Dacosta E, Kagina BM, Olivier J. Health systems constraints and facilitators of human papillomavirus immunization programmes in sub-Saharan Africa: a systematic review. Health Policy Plan. 2020 Jul 1;35(6):701-717. doi: 10.1093/heapol/czaa017. PMID 32538437
- [Background] Devarapalli P, Labani S, Nagarjuna N, Panchal P, Asthana S. Barriers affecting uptake of cervical cancer screening in low and middle income countries: A systematic review. Indian J Cancer. 2018 Oct-Dec;55(4):318-326. doi: 10.4103/ijc.IJC_253_18. PMID 30829264
- [Background] Lim JN, Ojo AA. Barriers to utilisation of cervical cancer screening in Sub Sahara Africa: a systematic review. Eur J Cancer Care (Engl). 2017 Jan;26(1). doi: 10.1111/ecc.12444. Epub 2016 Feb 7. PMID 26853214
- [Background] McFarland DM, Gueldner SM, Mogobe KD. Integrated Review of Barriers to Cervical Cancer Screening in Sub-Saharan Africa. J Nurs Scholarsh. 2016 Sep;48(5):490-8. doi: 10.1111/jnu.12232. Epub 2016 Jul 19. PMID 27434871
- [Derived] Iwelunmor J, Wapmuk AE, Kokelu E, Ojo T, Olusanya O, Gbaja-Biamila T, Akinsolu FT, Musa AZ, Xian H, Abodunrin OR, Kalulu P, Obiorah A, Afadapa M, Obodoechina N, Nwaozuru U, Anikamadu O, Smith J, Azuogu BN, Ajenifuja K, Jia M, Bamogo A, Babatunde A, Ong JJ, Zhang L, Zou Z, Airhihenbuwa CO, Tucker JD, Ezechi OC. For girls and women (4GW) HPV RCT protocol: a crowdsourced, pragmatic stepped-wedge cluster randomized trial to improve uptake of HPV vaccination and screening among mother-daughter dyads in Nigeria. Implement Sci. 2025 May 1;20(1):18. doi: 10.1186/s13012-025-01428-5. PMID 40312377
- See also: Global strategy to accelerate the elimination of cervical cancer as a public health problem — http://www.who.int/publications/i/item/9789240014107